CLINICAL TRIAL: NCT07119554
Title: The Effect of Postpartum Contraceptive Method Counseling Based on Health Belief Model on Family Planning Attitudes and Intention to Use Contraceptives
Brief Title: The Effect of Postpartum Contraceptive Method Counselling on the Intention to Use Family Planning Methods
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Melike Dissiz, Associate Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulSBU-HHF-MD-01
Record Dates: First submitted 2025-08-05; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Contraceptive Counseling
Keywords: Postpartum; Regulation of fertility; Contraception; Motivational interviewing

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial using motivational interviewing in two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBM-Based Counselling Group (Experimental): Participants in this group will receive individual contraceptive counselling based on the Health Belief Model (HBM) from the first month after birth until the sixth month.
  Interventions: Behavioral: HBM-Based Postpartum Contraceptive Counselling
- Standard care group (No Intervention): Participants in this group will receive only routine care provided by health facilities, without any structured contraceptive counselling during the postpartum period.

INTERVENTIONS:
Behavioral: HBM-Based Postpartum Contraceptive Counselling — This intervention involves providing a structured, individual contraceptive counseling session based on the Health Belief Model (HBM) to women in the postpartum period.The session is delivered face-to-face, lasts approximately 30 to 45 minutes, and is structured around the core components of the HBM: perceived susceptibility, perceived severity, perceived benefits, perceived barriers, self-efficacy, and cues to action. The aim of the intervention is to improve attitudes toward family planning and increase the intention to use contraceptive methods.
  Arms: HBM-Based Counselling Group

SUMMARY:
With the acceleration of developments in health technology, changes have occurred in professional knowledge and practices, as well as in patient needs and expectations. These changes have also influenced the way nursing care is delivered, leading to a shift from traditionally applied training methods to more modern and technology-based education tools. These include telephone counseling, online and web-based counseling, and the use of models.

In recent years, the use of motivational interviewing techniques in providing counseling services has become increasingly common in the field of nursing and is considered an effective communication method. In light of this information, the aim of this study is to evaluate the effect of postpartum contraceptive counseling based on the Health Belief Model using motivational interviewing techniques, along with spousal participation, on women's attitudes toward family planning and their intention to use contraceptives.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of postpartum contraception counselling based on the health belief model on family planning attitudes and contraceptive method use intentions. The study was designed as a randomised controlled trial. The study population will consist of women who visited the postpartum ward at Zeynep Kâmil Women's and Children's Diseases Training and Research Hospital in Istanbul between March 2025 and November 2025. In the study, the sample size was calculated using the 'G. Power-3.1.9.2' programme at a 95% confidence level prior to the data collection phase. The study will evaluate the effect of motivational interviews based on the Health Belief Model on family planning attitudes and contraceptive use intentions. Accordingly, the scores from the 'Family Planning Attitude Scale' (difference between the intervention and control groups) used in Tavukçu's (2024) study were referenced for calculation (63). Accordingly, it was estimated that the minimum sample size required for 80% power at a significance level of 0.05 and an effect size of 0.794 would be 26 participants per group (total 52). Considering that a 20% loss may occur during the research process, the sample is planned to consist of 62 participants (intervention group = 31, control group = 31). Data collection will begin after the necessary institutional permission, ethics committee permission, and scale usage permissions have been obtained. A simple randomisation method will be used to randomly select individuals from the population and assign them to the intervention and control groups without bias. Volunteers who meet the inclusion criteria will be informed about the study and their consent will be obtained before randomisation. Using the computer-assisted https://www.random.org/integers/ programme, 31 participants will be assigned to the intervention group and 31 participants to the control group using a simple randomisation method.

ELIGIBILITY:
Inclusion Criteria:

* Women who volunteered to participate in the study,
* were 18 years of age or older,
* were primiparous,
* spoke Turkish,
* owned a smartphone,
* had no chronic illness or diagnosed mental or psychiatric illness, were included in the study.

Exclusion Criteria:

* Women whose partners have undergone or will undergo a vasectomy, and women who have chosen tubal ligation will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female gender
Enrollment: 62 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in attitudes toward family planning and contraceptive method use intention scale scores at 6 months | in the 6th months after birth
  Postpartum contraceptive method counseling provided through motivational interviewing based on the health belief model

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Hamidiye Institute of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided